CLINICAL TRIAL: NCT05530902
Title: Multidisciplinary Primary Rehabilitation Care for Patients With Chronic Musculoskeletal Pain
Acronym: MPRC_CMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Zilveren Kruis (Unknown); Zorgverzekeraar CZ (Other); Zorgverzekeraar Menzis (Unknown); Rotterdam University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC-2022-0289
Record Dates: First submitted 2022-07-14; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with musculoskeletal pain (Experimental): Patients with musculoskeletal pain
  Interventions: Other: Multidisciplinary Primary Rehabilitation Care

INTERVENTIONS:
Other: Multidisciplinary Primary Rehabilitation Care — As described by the Policy Regulation 'Innovation' (NZa). The MPRC is a structured treatment program following the biopsychosocial approach, aiming to optimize functioning and participation in CMP patients. The treatment program is provided by paramedical specialists and, in cases that are more complex, a rehabilitation physician will be involved. The program has a diagnostic phase, a treatment phase (6-12 weeks) and a follow-up (12 months).

SUMMARY:
Rationale: A great variability in treatment contents, ways of collaboration between healthcare professionals, and evaluation methods for the treatment in chronic musculoskeletal pain (CMP), exists. Currently, multidisciplinary diagnostics, pain education and treatment in primary care, in collaboration with secondary care, especially with a biopsychosocial approach, is barely or not organized for patients having CMP. Objective: The aim of this study is to gain insight into the feasibility, health care and societal costs, effects regarding the patients' functioning and participation and perceived quality of care of the multidisciplinary primary rehabilitation care (MPRC) for different organization structures.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain (CMP) occurs in 18% of the Dutch population and may cause severe problems in daily functioning of patients. In 10% of the Dutch population, these problems are a leading cause of chronic disability, which leads to a high personal burden.

This will lead to high societal and health care costs. Most of these costs (80-90%) are the result of societal burden, such as work absenteeism, work productivity loss, social benefits and costs as a result of required (in)formal support from third parties (e.g. domestic help). According to the RIVM, the health care costs for neck and back pain are estimated at 937 million euro in 2017. This represents 14% of the total healthcare costs for musculoskeletal and tissue complaints and 1% of the total health care costs in The Netherlands.

The World Health Organization states that two-thirds of all conditions that need rehabilitation services comes from musculoskeletal disorders. With an ageing and growing population, the number people with musculoskeletal disorders increases fast, which will lead to a rapid increase of societal and health care costs. To decrease these costs, multidisciplinary rehabilitation workforce should be available. It is shown that multidisciplinary rehabilitation services in primary care and between primary care and secondary or tertiary care can be efficient. However, a great variability in treatment contents, ways of collaboration between healthcare professionals, and evaluation methods for the treatment in CMP exists.

The Dutch national care standard for CMP proposes an inventory of the factors contributing the causes and maintenance of pain and its associated limitations in daily functioning and participation. These factors can be divided in biomedical, psychological and societal factors: the biopsychosocial model. Since treatments focusing on this model have positive effects on patient outcomes, the standard recommends a biopsychosocial approach in designing a treatment plan. Thereby, the stepped care principles have to be taken into account for the treatment of CMP patient. In stepped care, the intensity of professional care is pre-defined. The stepped care principles contain the four following levels of care:

Step 1: prevention and self-management; Step 2: Monodisciplinary diagnostics, pain education and treatment in primary care; Step 3: Multidisciplinary diagnostics, pain education and treatment in primary care in collaboration with secondary care; Step 4: Multidisciplinary diagnostics, pain education and treatment in secondary or third care.

A great variability in treatment contents, ways of collaboration between healthcare professionals, and evaluation methods for the treatment in chronic musculoskeletal pain (CMP), exists. Currently, multidisciplinary diagnostics, pain education and treatment in primary care, in collaboration with secondary care (step 3), especially with a biopsychosocial approach, is barely or not organized for patients having CMP. Receival of the right health care treatment, at the right moment can therefore be restricted.

Presently, only restricted evidence exists, concerning the effectiveness of multidisciplinary primary care for CMP patients. Therefore, the Dutch Healthcare Authority (NZa) initiated an Policy Regulation 'Innovation' for multidisciplinary primary care. This study aims to gain insight into the feasibility, health care and societal costs, effects regarding the patients' functioning and participation and perceived quality of care of the multidisciplinary primary rehabilitation care (MPRC) for different organization structures.

Aims and hypotheses

The aim of this study is to gain insight into the feasibility, health care and societal costs, effects regarding the patients' functioning and participation and perceived quality of care of the multidisciplinary primary rehabilitation care (MPRC) for different organization structures. The research aims of this study are:

1. To evaluate the changes in functioning and participation of patients with CMP receiving MPRC, directly after the treatment, after six months follow-up and after 12 months follow-up as compared to baseline.
2. To evaluate the clinical relevance changes in functioning and participation of patients with CMP receiving MPRC, directly after the treatment, after six months follow-up and after 12 months follow-up.
3. To evaluate whether the changes in functioning and participation of patients with CMP receiving MPRC, directly after the treatment, after six months follow-up and after 12 months follow-up, differs between the different regions where the treatment is received.
4. To evaluate which prognostic factors may predict the level of changes in functioning and/or participation in CMP patients receiving MPRC after six months follow-up and after 12 months follow-up.
5. To evaluate the changes in (direct and indirect) costs for CMP patients receiving MPRC, post treatment compared to pretreatment.
6. To evaluate the feasibility of MPRC for patients with CMP.
7. To study the experiences of patients with CMP receiving MPRC.
8. To study the experiences of the healthcare professionals participating in the MPRC program for CMP patients.

Methodological approach

This study is a mixed-methods, multicenter study that will be conducted five local networks / health care settings in the Netherlands. The study will be conducted from May 2022 until August 2024. The health care settings participating this study offer their own developed treatment program to patients in its region. An independent research team will evaluate the effect of programs.

Study 1

Study design

1. The main field of study is a quantitative longitudinal cohort study whereby participating patients are asked to fill in a set of eight questionnaires. The set of questionnaires will be partly sent by the health care organizations and partly by the research group Study parameters Main study parameters are the perceived disability, measured with the Pain Disability Index (PDI) and the physical quality of life, measured with the Physical Component Scale (PCS) of the SF-12. Secondary study parameters are the mental quality of life (SF-12), health-related productivity losses (iPCQ), health care consumption (iMCQ), work ability (WAS), self efficacy (PSEQ), life participation: (USER-P ggz), anxiety and depression (HADS), catastrophizing (PCS-6), satisfaction with care (PREM) and complexity of musculoskeletal problems (STarT MSK tool).

   Study procedures The patients participating the study will be asked to complete a set of eight questionnaires at the start of the treatment, the diagnostic phase/intake (T0), after the intensive treatment phase, three months after T0 (T1); after the intensive treatment phase, nine months after T0 (T2) and after the intensive treatment phase, fifteen months after T0 (T3). The set of questionnaires will partly be sent by the health care settings and partly by the research group. These questionnaires are provided electronically (the EPD-system of the health care setting, Castor EDC and LDOT). On request, a paper-version of the set of questionnaires can be provided. The results will be used by the health care professional to determine the treatment plan, to assess the effect of the treatment and a adjust the treatment plan based on the patients' current needs.

   Study 2 and 3 Study design
2. Evaluation on the feasibility of the treatment and the organization of the MER will be executed. Data on this subject will be collected via the Electronic Patient Dossier of the health care settings
3. Two qualitative focus group studies will be performed on the experiences and satisfaction with the MER from both the perspective of the health care professionals and the participating patients Study parameters The following prognostic data and patient selection data will be collected: patient characteristics, physical and psychiatric co-morbidity, duration of current complaint episodes, complicating physical or social factors, perceived social support, treatment received in the last year, recidivism and received help when filling in the questionnaires

Study procedures Qualitative research Three months after the intensive treatment phase a random selection of participating patients will be invited to participate in a phone interview. Topics that will be addressed are related to the content of the treatment, satisfaction with the treatment, history of the pain complaints, history of health care consumption and improvement recommendations. Furthermore, participating health care professionals will be invited to participate in an online focus group interview per health care setting. The focus group interviews will take place at the start of the project, after six months after the start of the project and after 18 months after the start of the project. Topics that will be addressed are related to the professionals satisfaction with the M, the process of the MPRC and the feasibility of the MPRC.

Feasibility The participating health care professionals will be asked to collect and deliver the following patient data to the research team, which will be used for the process evaluation: healthcare professionals' disciplines that are involved in the treatment program, the amount of treatment sessions, frequency and content of healthcare professionals' collaboration, (frequency of) coordination, communication and collaboration with general practitioners, patients' adherence and planning, executing and declaring the MPRC. Besides that, the following data will be collected and analyzed: compliance, feasibility and duration of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* musculoskeletal pain
* duration of musculoskeletal pain ≥ 3 months
* monodisciplinary primary care is completed

Exclusion Criteria:

* previous experiences with treatment in multidisciplinary secondary or tertiary care
* Co-morbidities limiting to complete the treatment program within the preset time
* BMI ≥ 35
* present addiction or other psychiatric problems
* inadequate understanding of the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes in perceived level of disability | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  Measured with the Pain Disability Index (PDI) questionnaire
Changes in physical quality of life | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  Measured with the Physical Component Scale (PCS) of the SF-12 questionnaire

SECONDARY OUTCOMES:
Changes in health-related productivity losses | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  Measured with the iMTA Productivity Cost Questionnaire (iPCQ) Questionnaire (iPC)
Changes in health care consumption | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  Measured with the iMTA Medical Consumption Questionnaire (iMCQ)
Changes in work ability | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  Measured with the Work Ability score (WAS) questionnaire.
Changes in self efficacy | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  Measured with the Pain Self Efficacy Questionnaire (PSEQ)
Changes in life participation | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  Measured with the USER-Participation (USER-P)
Changes in anxiety and depression | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  Measured with the Hospital Anxiety and Depression Scale (HADS)
Changes in catastrophizing | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  Measured with the Pain Catastrophizing Scale (PCS)
Changes in satisfaction with care | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  Measured with the Patient Reported Experience Measure' (PREM)
Changes in complexity of musculoskeletal problems | At the start of the treatment (the diagnostic phase) (T0), at three months (T1); at nine months (T2) and at fifteen months (T3).
  STarT MSK tool

CONTACTS AND LOCATIONS:
Locations (5):
- Netherlands (5):
  - OCA, Eindhoven
  - Activos, Goes
  - Belife, Rotterdam
  - Eenplus, Velp
  - CIR, Zwolle

IPD SHARING:
Plan to Share IPD: No